CLINICAL TRIAL: NCT03591315
Title: Multimodal Evaluation on Visual Pathway Predicts the Surgical Curative Effects in Sellar Area Tumors
Brief Title: Clinical Study of Structural and Functional Evaluation of the Visual Pathway
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 201611627
Record Dates: First submitted 2018-06-21; First posted 2018-07-19 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-06

CONDITIONS: Pituitary Adenoma; Visual Impairment; Sellar Tumor; Neuroimaging
Keywords: visual pathway; functional magnetic resonance imaging; pituitary adenoma
MeSH Terms: conditions — Pituitary Neoplasms; Vision Disorders | interventions — Diffusion Tensor Imaging; Visual Field Tests; Visual Acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TG group: Patients with visual impairment caused by chiasma compression from sellar area tumors will undergo the following examinations: resting state fMRI, visual tasking state fMRI, diffusion tensor imaging (DTI), visual acuity and automated visual field test.
  Interventions: Diagnostic Test: resting state fMRI; Diagnostic Test: visual tasking state fMRI; Diagnostic Test: diffusion tensor imaging; Diagnostic Test: automated visual field; Diagnostic Test: visual acuity
- HC group: Volunteers with no visual impairment(visual acuity of both eyes >1.0) or Nervous System disease will undergo the following examinations: resting state fMRI, visual tasking state fMRI, diffusion tensor imaging (DTI), visual acuity and automated visual field test.
  Interventions: Diagnostic Test: resting state fMRI; Diagnostic Test: visual tasking state fMRI; Diagnostic Test: diffusion tensor imaging; Diagnostic Test: automated visual field; Diagnostic Test: visual acuity

INTERVENTIONS:
Diagnostic Test: resting state fMRI — Define the visual resting state network.
  Other Names: V-RS
Diagnostic Test: visual tasking state fMRI — Using visual task stimulation to identify the activation characteristic of primary visual cortex.
Diagnostic Test: diffusion tensor imaging — Define the integrity of white matter fibers in the visual pathway.
  Other Names: DTI
Diagnostic Test: automated visual field — Identify the existence and type of visual field defect.
  Other Names: VF
Diagnostic Test: visual acuity — Assess the visual acuity by using ETDRS scales.
  Other Names: VA

SUMMARY:
Sellar area tumors such as pituitary adenoma, craniopharyngioma and meningioma, etc, commonly lead to visual impairment symptoms. Patients suffer from a loss of visual acuity (VA) and visual field defects (VF) due to a local compression on the optic chiasma by the tumor. In the management of these patients, it is an important goal to evaluate their visual function throughout the treatment, so as to predict the outcome of the visual function .

Since the visual pathway contains a huge complex network of both structure and function, traditional simplex evaluation of VA and VF is obviously not enough. Former studies have revealed changes in the visual network and cortex structure in neurodegenerative diseases and optic neuritis, yet the functional and structural changes caused by local tumor compression and their relation to the visual cortex activity patterns needs further research.

The objective of this research is to asses the visual function in patients with sellar area tumor 1 week preoperatively (baseline),72 hours postoperatively(checking point 1) and at 3 months follow up(checkpoint 2). By using multimodal evaluation including visual resting and task state fMRI, diffusion tensor imaging (DTI), etc. The investigators aim to reveal the changes in functional connectivity (FC), amplitude of low frequency fluctuation (ALFF), regional homogeneity (REHO) ,visual cortex activity patterns and tract-based spatial statistics (TBSS).

DETAILED DESCRIPTION:
Detailed Description:

Study objective

Visual pathway contains both structural and functional network. When it is impacted by neurodegenerative diseases, neuritis or direct mechanical pressure, visual impairment occurs due to damage to the pathway. Former study on Parkinson's disease (Dagmar H. Heep et al, Radiology, 2017 ) found loss of functional connectivity in posterior and paracentral brain regions, while a study on optic neuritis (Yael Backner et al, JAMA Neurology,2018) showed an increase in functional connectivity and slightly loss in optic fiber integrity. Instead of simplex resting-state fMRI，the investigators of this study aim to assess:

1. whether similar changes in functional networking occur when visual pathway is impacted by chiasma compression from tumors in sellar area (by resting-state fMRI).
2. The correlation between local chiasma compression and visual cortex activation pattern ( by visual tasking-state fMRI).
3. Changes and recovery of the white matter fiber structure in the visual pathway.

( by diffusion tensor imaging, DTI).

Method Participants: 60 adult participants (18-60 years old ) will be enrolled in the department of Neurosurgery at Xiangya Hospital of Central South University. The experimental arm will consist of 30 patients with visual impairment symptoms caused by chiasma compression by sellar area tumors (Tumor Group, TG). The control arm will consist of 30 healthy controls without any nervous system disease or visual impairment (Healthy Control Group, HC, control arm).

Study design: Transversal and Longitudinal, single center, comparative study is designed to evaluate functional and structural visual networking of sellar area tumor patients and healthy controls. The study involves assessment with resting-state fMRI, tasking-state fMRI and DTI. Patients of experimental arm will be evaluated by multimodal fMRI at 3 different checkpoints (baseline is 1 week preoperative ,checkpoint 1 is 72 hours postoperative ,checkpoint 2 is 3 months follow up ). Participants of control arm will be evaluated only once. Transversal comparison will be conducted between preoperative tumor patients and healthy controls, while longitudinal comparison will be within tumor group at baseline and two other different checkpoints.

MRI data acquisition and analysis strategy: In this study, the MRI data is acquired by Siemens 3.0T Prisma scanner, including sequences of mprage T1 , diffusion tensor imaging, resting-state fMRI and visual stimulation task fMRI. Resting-state fMRI longitudinal data analysis includes functional connectivity (FC), amplitude of low frequency fluctuation (ALFF) and regional homogeneity (REHO) to assess visual functional networking in both group. These Data wil be analysed using a multivariate approach and independent component analysis (ICA). Visual tasking fMRI will be conducted under classic black and white "chess board" simulation on each eye. For the evaluation of structural visual network, afferent visual pathway (optic tract and radiation ), fiber tracking as well as tract-based spatial statistics (TBSS) will be analyzed within both arms at baseline,checkpoint 1 and checkpoint 2 of the experimental arm will verify changing and recovering process of the visual pathway after chiasma decompression.

Primary outcomes

1. The difference in visual pathway anatomy and functional network between preoperative sellar area tumor patients and healthy controls. Tumor patients will be evaluated clinically by visual acuity (VA), visual field (VF), tumor height and chiasma thickness.
2. The verification of the correlation between patterns of chiasma compression and visual cortex activity. Revealing the difference of visual cortex activity patterns between both arms.

Secondary outcomes Throughout the 3 months follow up of the experimental arm patients, observe and verify the recovery process of both functional and structural visual network after chiasma decompression and evaluate its correlation with clinical visual function outcome.

Statistics

1. An analysis of two sample T test between the two groups will be performed to assess the difference of FC,REHO,ALFF and visual cortex activity pattern between resting state data and data from the visual task of TG and HC.
2. An analysis of variance (ANOVA) within TG group will be performed to assess the changes and recovery of FC, REHO, ALFF and visual cortex activity pattern via resting state data and data from the visual task's data.

Correlations will be explored between multimodal fMRI parameters (both functional and structural) and clinical criteria (e.g VA,VF, tumor size, visual outcome, etc).

ELIGIBILITY:
Inclusion Criteria:

1. patients with sellar area tumors ( including pituitary adenoma,craniopharyngioma and meningioma) resulting a visual deficit (loss of visual acuity or visual field).
2. Male or female between 18y to 60y.
3. Patients treated with transsphenoidal surgery.
4. Patients agreeing to participate in the study and willing to sign an informed consent.

Exclusion Criteria:

1. tumor height ≥ 4cm.
2. Patients with recurrent tumors, previous craniotomy or gamma knife treatment
3. Visual impairment caused by other diseases.
4. Mental disorders, inability to cooperate with treatment and follow up visits.
5. Patients with other serious complications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Admitted sellar area tumor patients in the Neurosurgery Department at Xiangya Hospital of Central South University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change on functional connectivity of visual resting network | Change from baseline (1 week preoperative) functional connectivity of visual resting network at 3 days postoperative and 3 moths postoperative.
  Outcomes of visual resting state fMRI to assess the functional connectivity (FC) of visual resting network.
Change on signal strength of the visual cortex activation by visual tasking state fMRI (visual BOLD fMRI). | Change from baseline (1 week preoperative) visual cortex activation signal strength at 3 days postoperative and 3 moths postoperative.
  Outcomes of visual BOLD fMRI to assess the function of visual cortex by measuring the signal strength (T-test score) of the visual cortex activation.
Change on anatomical Connectivity of the posterior visual pathway | Change from baseline (1 week preoperative) TBSS result at 3 days postoperative and 3 moths postoperative.
  Outcomes of tract-based spatial statistics (TBSS) to assess the integrity of the white matter fibers in the posterior visual pathway.

SECONDARY OUTCOMES:
Change on visual acuity | Change from baseline (1 week preoperative) visual acuity at 3 days postoperative and 3 moths postoperative.
  Outcomes of visual acuity test for evaluation of the visual function impairment and recovery.
Change on visual field. | Change from baseline (1 week preoperative) visual field at 3 days postoperative and 3 moths postoperative.
  Visual Field Defects via Humphrey visual field chart, Mean Deviation and Standard Deviation in the patients' group at different checkpoints.
Change on amplitude of low frequency fluctuation (ALFF) of visual resting network | Change from baseline (1 week preoperative) ALFF of visual resting network at 3 days postoperative and 3 moths postoperative.
  Visual resting state fMRI data will be analysed to assess the ALFF data of visual resting network
Change on regional homogeneity (REHO) of visual resting network | Change from baseline (1 week preoperative) REHO of visual resting network at 3 days postoperative and 3 moths postoperative.
  Outcomes of visual resting state fMRI to assess the regional homogeneity (REHO) of visual resting network.
Change on fractional atrophy (FA) value of the posterior visual pathway. | Change from baseline (1 week preoperative) FA of the posterior visual pathway at 3 days postoperative and 3 moths postoperative..
  Outcomes of fractional atrophy (FA) on the posterior visual pathway via diffusion tensor imaging (DTI) and fiber tractography.
Change on axial diffusivity (AD) of the posterior visual pathway. | Change from baseline (1 week preoperative) AD value of the posterior visual pathway at 3 days postoperative and 3 moths postoperative..
  Outcomes of axial diffusivity (AD) value on the posterior visual pathway via diffusion tensor imaging (DTI) and fiber tractography.
Change on radial diffusivity (RD) of the posterior visual pathway. | Change from baseline (1 week preoperative) RD value of the posterior visual pathway at 3 days postoperative and 3 moths postoperative..
  Outcomes of radial diffusivity (RD) value on the posterior visual pathway via diffusion tensor imaging (DTI) and fiber tractography.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Z Xiong, MD/PhD, Study Chair — Neurosurgery department, Xiangya Hospital of Central South University, Changsha, Hunan, China
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Backner Y, Kuchling J, Massarwa S, Oberwahrenbrock T, Finke C, Bellmann-Strobl J, Ruprecht K, Brandt AU, Zimmermann H, Raz N, Paul F, Levin N. Anatomical Wiring and Functional Networking Changes in the Visual System Following Optic Neuritis. JAMA Neurol. 2018 Mar 1;75(3):287-295. doi: 10.1001/jamaneurol.2017.3880. PMID 29297053
- [Result] Hepp DH, Foncke EMJ, Olde Dubbelink KTE, van de Berg WDJ, Berendse HW, Schoonheim MM. Loss of Functional Connectivity in Patients with Parkinson Disease and Visual Hallucinations. Radiology. 2017 Dec;285(3):896-903. doi: 10.1148/radiol.2017170438. Epub 2017 Sep 27. PMID 28952907